CLINICAL TRIAL: NCT02738528
Title: APPLICATION OF MENTAL PRACTICE IN MOTOR LEARNING OF BRUSHING ON PEOPLE WITH PARKINSON
Brief Title: MENTAL PRACTICE IN MOTOR LEARNING OF BRUSHING AND PARKINSON DISEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, CARLA CABRAL DOS SANTOS ACCIOLY LINS, PhD PRINCIPAL INVESTIGATOR, Universidade Federal de Pernambuco
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE N°. 29242414.2.0000.5208
Record Dates: First submitted 2016-04-08; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): Mental practice and brushing guidance in patients with Parkinson Disease
  Interventions: Other: Mental practice and brushing guidance in patients with Parkinson Disease
- Control group (No Intervention): Brushing guidance in patients without Parkinson Disease

INTERVENTIONS:
Other: Mental practice and brushing guidance in patients with Parkinson Disease
  Arms: Experimental Group

SUMMARY:
Parkinson's disease (PD) is characterized by dopaminergic neurons degeneration of the substantia nigra, in the midbrain, resulting in the presence of motor disorders, such as tremor, rigidity, bradykinesia, and postural instability. Researches have shown that mental rehearsal in learning motor skills through mental practice (MP), which associates the physical practice to somatosensory imagination to action, causes positive effects in several motor tasks, such as the speed of motion, muscle strength performance and accuracy. Thus, this study aims to report the effects of MP as a tooth brushing training strategy in people with Parkinson's disease. This project was approved by the Ethics Committee in Research with Human beings of UFPE and attempt to compare the presence of bacterial biofilm before and after 8 weeks of brushing through the mental practice training, based on O'Leary's index. The sample consisted of 35 people, divided into two groups: Intervention Group consists of 17 people with Parkinson's, in stages I to III of the disease, who underwent brushing orientation associated with PM, and the control group people without the disease, who received only orientation brushing. Then, the data were evaluated by factorial ANOVA 2x2 and post hoc Tukey test considering p <0.05. It was observed that after the intervention was a significant improvement of the control dental biofilm.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80 years;
* Idiopathic PD Clinical Diagnostics according to the Bank of brain London;
* Patients in stages I to III according to Hoehn and Yahr;
* Satisfactory communicative and cognitive level checked by the Mini-Mental State Examination;
* Subject to satisfactory clinical, lying in his home in the care of relatives;
* Patients who possessed a sextant of the dental arch with teeth.

In the control group individuals without neurological disease were included: both sexes at ages similar to the group with PD, satisfactory health, active life, and natural teeth.

Exclusion Criteria:

* Another neurological disease associated with PD;
* Mioarticulares abnormalities in the upper limbs to prevent their use for independent brushing;
* Use of orthotic / prosthetic hand;
* Toothless in both dental arches.

In the control group were excluded individuals with mioarticulares abnormalities of the upper limbs; in use of orthotic / prosthetic hand; presenting any movement disorder in the upper limbs.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Dental biofilm | 8 weeks
  Based on O'Leary's index, the calculation was made dividing the number of surfaces stained by the total number of scanned surfaces, multiplied by 100.

IPD SHARING:
Plan to Share IPD: No